CLINICAL TRIAL: NCT03063359
Title: Non-inferiority of Intranasal Fentanyl Versus Oral Morphine Sulfate in the Treatment of Pain in Pediatric Trauma : a Controled Randomized , Single Blind Study
Brief Title: Intranasal Fentanyl Versus Oral Morphine Sulfate in the Treatment of Pain in Pediatric Trauma
Acronym: FINDOL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The new pain protocols imposed by the HAS make it difficult to include new patients in the study
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9732
Record Dates: First submitted 2017-01-30; First posted 2017-02-24 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Pain, Acute
Keywords: traumatic pain; children; fentanyl; intranasal use
MeSH Terms: conditions — Acute Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal fentanyl + Oral placebo (Experimental): Administration of intranasal fentanyl (1.5µg/kg) and oral placebo in children with acute pain in traumatic context on arrival in emergency pediatric department.
  Interventions: Drug: Intranasal fentanyl + Oral Placebo
- Oral morphine + Intranasal placebo (Active Comparator): Administration of oral morphine (0.4mg/kg) and intranasal placebo in children with acute pain in traumatic context on arrival in emergency pediatric department.
  Interventions: Drug: Oral Morphine + Intranasal Placebo

INTERVENTIONS:
Drug: Intranasal fentanyl + Oral Placebo — Administration of intranasal fentanyl (1.5µg/kg) and Oral placebo (NaCl 0.9%) in children with acute pain in traumatic context on arrival in emergency pediatric department.
  Other Names: Intranasal Fentanyl + Oral NaCl
  Arms: Intranasal fentanyl + Oral placebo
Drug: Oral Morphine + Intranasal Placebo — Administration of oral morphine (0,4mg/kg) and intranasal placebo (NaCl 0.9%) in children with acute pain in traumatic context on arrival in emergency pediatric department.
  Other Names: Oral Morphine + Intranasal NaCl
  Arms: Oral morphine + Intranasal placebo

SUMMARY:
Acute tramatic pain is one of main reasons for consultation in pediatric emergency departments.

To manage pain quickly and effectively must be a primary outcome of the emergency department. However, pediatric emergency department are sometimes criticized for inadequate and delayed initiation analgesia . Indeed, several studies have shown the inadequacy between the intensity of the pain evaluated by the care team and the therapeutic management of it.

The ideal analgesic must have a rapid onset of action, have a powerful analgesic effect, have few side effects and can be administered quickly and painlessly. That's why, the main outcome of this study is to assess the non inferiority of a treatment by intranasal Fentanyl vs morphine sulfate (oral use) in children with traumatic pain on arrival to pediatric emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 4 years old and 15,3 years old
* Acute pain in traumatic context with a suspicion of fracture for patient <7years old : feeling Pain >6/10 defined with a face analogue scale and a visual analogic scale (the difference between the scales is not <10 points)
* For patients >7 years old : feeling pain >6 points and defined thanks to a visual analogic scale
* Informed consent form signed by parents
* Beneficiary of an european health protection

Exclusion Criteria:

* Antalgic ( II or III) within 4 hours before the inclusion
* Allergic or non-indication of fentanyl
* Allergic or contraindication of morphine sulfate
* Pre existing peripheral intravenous catheter
* Traumatic brain injury
* Nasal traumatic

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Assessment of the value of the pain feeling | 45 minutes
  Assessment of the value of the pain feeling measured by visual analogic scale

SECONDARY OUTCOMES:
Delay in treatment efficacy | up to 45 minutes
  Delay in treatment efficacy measured by a reduction of pain (1 point) assessed by visual analogic scale from the administration of the treatement.

CONTACTS AND LOCATIONS:
Overall Officials: Gaël GG GUYON, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided